CLINICAL TRIAL: NCT06485388
Title: The Effects of Propofol and Thiopental on Nitric Oxide Production and Release in Erythrocytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melike Cengiz (Other)
Responsible Party: Sponsor-Investigator, Melike Cengiz, MD,Professor Doctor, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Akdeniz U. Faculty
Record Dates: First submitted 2024-03-17; First posted 2024-07-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Effect of Drug
Keywords: nitric oxide; erythrocyte; propofol; thiopental
MeSH Terms: interventions — Propofol; Thiopental

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiopental (Active Comparator): Venous blood samples will be taken from the patients included in the study and incubated with thiopental (dose: 100, 250, 500 and 1000µM) after appropriate procedures in the laboratory environment. . After incubation, all resuspensions will be subjected to flow cytometric analysis to evaluate erythrocyte NO synthase activity and erythrocyte-mediated NO release.
  Interventions: Drug: Thiopental
- Propofol (Active Comparator): Venous blood samples will be taken from the patients included in the study and incubated with propofol (dose: 100, 250, 500 and 1000µM) after appropriate procedures in the laboratory environment. . After incubation, all resuspensions will be subjected to flow cytometric analysis to evaluate erythrocyte NO synthase activity and erythrocyte-mediated NO release.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Venous blood samples will be taken from the patients included in the study and incubated with propofol (dose: 100, 250, 500 and 1000µM) after appropriate procedures in the laboratory environment. . After incubation, all resuspensions will be subjected to flow cytometric analysis to evaluate erythrocyte NO synthase activity and erythrocyte-mediated NO release.
  Arms: Propofol
Drug: Thiopental — Venous blood samples will be taken from the patients included in the study and incubated with thiopental (dose: 100, 250, 500 and 1000µM) after appropriate procedures in the laboratory environment. . After incubation, all resuspensions will be subjected to flow cytometric analysis to evaluate erythrocyte NO synthase activity and erythrocyte-mediated NO release.
  Arms: Thiopental

SUMMARY:
Hypotension is frequently encountered during the use of these commonly used intravenous anaesthetic agents (thiopental and propofol). This is thought to be a consequence of their effects on the sympathetic nervous system, myocardial contractility or vascular tone. However, propofol causes a greater fall in systemic arterial blood pressure than any other drug used for induction of anaesthesia. Propofol causes profound vasodilation, whereas its myocardial depressant effect is not clear. The vasodilatation occurs in both arterial and venous systems. The decrease in systemic arterial blood pressure after thiopental induction is mainly due to peripheral vasodilatation caused by depression of the medullary vasomotor centre and inhibition of the sympathetic nervous system. However, how this peripheral vasodilator effect occurs after both drugs and which mediators accompany it have not yet been fully elucidated. In previous studies, it has been emphasised that systemic vasodilation may be related with increased formation of nitric oxide (NO), a small gaseous and lipophilic molecule which plays an important role in the regulation of vascular homeostasis and haemoregulation. It is important to elucidate the mechanisms that may mediate thiopental- and propofol-mediated vasodilatation in future studies in order to help the methods and treatments that can be developed to prevent hypotension caused by these drugs, which are widely used in clinical practice. Therefore, the aim of this study was to investigate the effects of thiopental and profol on erythrocyte NO synthase activity and erythrocyte-mediated NO release.

DETAILED DESCRIPTION:
Male patients aged 18-45 years with ASA (American Society of Anaesthesiologists) class I (normal, healthy person without any disease or systemic problem other than surgical pathology that does not cause a systemic disorder) who applied to the anaesthesiology and reanimation clinic outpatient clinic for preoperative preparation were planned to be included in the study. Women, patients with ASA class >1, patients with known thiopental/propofol allergy and patients outside the age range of 18-45 years were excluded from the study. Venous blood samples will be taken from the patients included in the study and incubated with thiopental and propofol (dose: 100, 250, 500 and 1000µM) after appropriate procedures in the laboratory environment. . After incubation, all resuspensions will be subjected to flow cytometric analysis to evaluate erythrocyte NO synthase activity and erythrocyte-mediated NO release.All patients included in the study will be informed and their written and verbal consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* Aged 18-45 years
* ASA (American Society of Anaesthesiologists) class I (normal, healthy person without any disease or systemic problem other than surgical pathology that does not cause a systemic disorder)

Exclusion Criteria:

* Women patients
* ASA class >1
* Patients with known thiopental/propofol allergy
* Patients outside the age range of 18-45 years

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
The effects of thiopental and propofol on erythrocyte NO synthase activity and erythrocyte-mediated NO release. | 120 days
  Blood samples will be taken from healthy human volunteers aged 25-45 years. Measurements will be performed using the fluorescent NO probe 4-amino-5-methylamino-20,70-difluorofluorescein diacetate. Propofol and thiopental will be added to the suspensions at doses of 100, 250, 500 and 1000 µM and incubated for 30 minutes. We will repeate these experiments in the presence of L-NAME, a non-specific nitric oxide synthase inhibitor. The nitrite/nitrate concentration will be measured in the supernatant of the erythrocyte suspensions after centrifugation.Intracellular calcium measurements will also be made during propofol and thiopental experiments. Fluo-4 calcium dye will be added to the medium and flow cytometric measurements will be repeated.

SECONDARY OUTCOMES:
The effects of thiopental and propofol on erythrocyte haemorheology | 120 days
  The effects of thiopental and propofol on erythrocyte haemorheology. Blood samples will be taken from healthy male volunteers and leucocytes will be extracted. The RBC deformability will be measured as an elongation index (EI) for various liquid shear stresses by laser diffraction analysis using an ectacytometer (LORRCA, RR Mechatronics, Hoorn, The Netherlands).RBC aggregation will be assessed using the same echacytometer. Aggregation will be determined by placing 1 ml of blood in the space between the cup and bob. The sample will then be sheared at a speed of 800 1/s for 10 seconds to disperse pre-existing aggregates. After 10 seconds, the shear will be abruptly reduced to zero and the level of laser light reflected from the sample will be digitally recorded for 120 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Arslan Yildiz, MD, Principal Investigator — Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey; Pinar Ulker, PhD, Principal Investigator — Akdeniz University School of Medicine, Department of Physiology; Ahmet Yildirim, Principal Investigator — Akdeniz University School of Medicine, Department of Physiology; Ayse Gulbin Arici, Professor, Principal Investigator — Akdeniz University School of Medicine, Department of Anesthesiology and Reanimation, Turkey; Murat Yilmaz, Professor, Principal Investigator — Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey
Locations (1):
- Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No